CLINICAL TRIAL: NCT05698017
Title: Phase 1 Open-Label Study for Treatment of Early to Moderate Stage Multiple System Atrophy Patients With the Investigational Allogeneic Cell Therapy Product, hOMSC300
Brief Title: Study to Evaluate Investigational Allogeneic Cell Therapy Product hOMSC300 for Treatment of Early to Moderate Stage Multiple System Atrophy (MSA)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cytora Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Cyt MSA hOMSC300
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Multiple System Atrophy; MSA - Multiple System Atrophy
Keywords: multiple system atrophy; MSA; stem cells; intrathecal
MeSH Terms: conditions — Multiple System Atrophy; Shy-Drager Syndrome

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to one of the following arms:
  1. The first 2 subjects recruited will be treated with the Low dose single Intrathecal (IT) administration of hOMSC300
  2. The following 2 subjects recruited will be treated with the High dose single intrathecal (IT) administration of hOMSC300; In the absence of any treatment related SAEs, the remaining patients (6) will be treated with the high dose, without further staggering.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose hOMSC300 (Experimental): Single IT administration of low dose hOMSC300
  Interventions: Biological: hOMSC300
- High dose hOMSC300 (Experimental): Single IT administration of high dose hOMSC300
  Interventions: Biological: hOMSC300

INTERVENTIONS:
Biological: hOMSC300 — Human Oral Mucosa Stem Cells

SUMMARY:
Purpose of this phase 1 study is to assess the safety of intrathecal administration of allogeneic human oral mucosa stem cells (hOMSCs) in patients suffering from early to moderate stage Multiple System Atrophy (MSA)

ELIGIBILITY:
Inclusion Criteria:

* Patient was diagnosed with probable MSA-C (cerebellar) or MSA-P (parkinsonian) variant within 60 months of symptom onset (excluding impotence)
* Subject can ambulate without the assistance of another person, defined as the ability to take at least 10 steps. Use of assistive devices is allowed
* Patient cognitive state permits him to sign informed consent, according to the PI's clinical judgement, and MoCA >= 24

Exclusion Criteria:

* Pregnant women and women before menopause
* Participants with a clinically significant or unstable medical or surgical condition that, in the opinion of the investigator, might preclude safe completion of the treatment or affect the treatment outcome.
* Patients with thrombocytopenia, other bleeding diathesis or taking anticoagulant therapy (not including Aspirin up to 100mg per day)
* Patients with known hypersensitivities to Plasmalyte, Gadolinium, Penicillin, and with general hypersensitivity to antibiotics
* Patients who fulfill the criteria of Parkinson's Disease
* History of electroconvulsive therapy
* History of brain surgery

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-02-19 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment related serious adverse events (SAEs) | 18 months
Number of participants with treatment related adverse events (AEs) | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Sourasky Medical Center (Ichilov), Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No